CLINICAL TRIAL: NCT01597440
Title: Long-term Outcome of N-Carbamylglutamate Treatment in Propionic Acidemia and Methylmalonic Acidemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Mendel Tuchman (Other)
Collaborators: Children's National Research Institute (Other); Boston Children's Hospital (Other); University Hospitals Cleveland Medical Center (Other); University of California, Los Angeles (Other); Children's Hospital of Philadelphia (Other); Lucile Packard Children's Hospital (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Mendel Tuchman, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCGC 0007
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Propionic Acidemia; Methylmalonic Acidemia
Keywords: Propionic acidemia (PA); Methylmalonic acidemia (MMA); Carbaglu NCG; Hyperammonia
MeSH Terms: conditions — Propionic Acidemia; Methylmalonic acidemia | interventions — N-carbamylglutamate; carglumic acid; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Carbamylglutamate (Experimental): Active NCG & Standard of Care
  Interventions: Drug: N-carbamylglutamate; Other: Standard of Care
- Placebo (Placebo Comparator): Standard of Care therapy
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: N-carbamylglutamate — Active NCG & Standard of Care Chemical Composition: N-carbamyl-L-glutamic acid (NCG) The daily dose will be 100 mg/kg/ day. The doses are to be divided into 2 equal doses and administered orally or enterally by nasogastric or gastrostomy tube (standard of care will prevail when choosing the mode of drug administration).
  The tablets must be dispersed in a minimum of 2.5-10 ml of water and ingested immediately or administered by fast push through a syringe via a nasogastric or gastrostomy tube. The suspension has a slightly acidic taste.
  This drug will be administered for 7 days after admission or until discharge (whichever is sooner).
  Other Names: Carbaglu; NCG
  Arms: N-Carbamylglutamate
Other: Standard of Care — Standard of Care

SUMMARY:
Background: Very few drugs exist that treat hyperammonemia, specifically PA and MMA. Diet restrictions and alternate pathway agents are the current primary treatments, but they frequently fail to prohibit brain damage.

Orthotopic liver transplantation cures the hyperammonemia of urea cycle disorders, but organ availability is limited and the procedure is highly invasive and requires life-long immunosuppression.

A drug that could repair or stimulate a dysfunctional urea cycle such as this would have several advantages over current therapy. A drug called N-carbamyl-L-glutamate, Carglumic acid (NCG or Carbaglu)has recently been found to be virtually curative of another urea cycle defect called NAGS deficiency. In this disorder, treatment with NCG alone normalizes ureagenesis, blood ammonia and glutamine levels, allows normal protein tolerance and restores health. Knowledge from this study is being applied to acquired hyperammonemia, specifically in patients with propionic PA and MMA, to try and improve neurodevelopmental outcomes by improving the hyperammonemia.

Aims: The overall objective of this project is to determine whether treatment of acute hyperammonemia with Carglumic acid in propionic acidemia (PA), methylmalonic acidemia (MMA) changes the long-term outcome of disease and to determine if it is effective in restoring urine ammonia levels to normal levels.

DETAILED DESCRIPTION:
Methods/Design This 5-year, Phase II, double-blind study aims to recruit and enroll 34 PA and MMA patients during acute episodes of hyperammonemia.

The primary aim is to circumvent the long-term neurodevelopmental decline due to having a prolonged levels of ammonia during crisis in the blood and urine. After treatment and crisis resolution with Carbaglu or placebo and standard of care therapy, measures of neurodevelopmental outcomes (Bayley II and Functional Status Scale) are being measured at 9, 15,21 and 30 months post-discharge from the hospital. Safety of NCG treatment will also be monitored as measured by close examination of adverse events and laboratory blood tests. To test for the effectiveness of NCG, longitudinal models to evaluate the groupwise difference (NCG vs. Placebo) in the trajectory of change in neurodevelopmental outcomes and safety analyses between drug and placebo patients.

Subsequent Episodes At any time after the initial episode, participants may present to the hospital with PA- or MMA-associated symptoms. If the plasma ammonia level verified as a bonafide episode of HA (plasma ammonia is ≥ 100 µmol/l), that participant will receive the same study medication that they received during their initial episode in a double-blinded fashion, (i.e. If the participant received NCG at the time of initial randomization, he/she will continue to receive NCG at each subsequent HA episode. If the participant received PLBO at the time of initial randomization, he/she will continue to receive PLBO at each subsequent HA episode). Only the pharmacist will know if the participant receives NCG or PLBO. The same study assessments (previously stated) will be conducted at each qualifying HSA episode.

ELIGIBILITY:
Inclusion Criteria

* Aged 4 weeks or younger (0-28 days)
* >36 weeks gestational age at birth
* Birth weight ≥2500 g
* Plasma ammonia level at presentation >150 mcmol/L
* PA or MMA presumed or established diagnosis as follows (one of the following):

  1. Acidosis at presentation, pH <7.3 OR
  2. Plasma acylcarnitine analysis either alone or as part of newborn screening, demonstrating C3 >4 mcmol/L OR
  3. Diagnosed, or sibling diagnosed with PA by semi-quantitative urine organic acid analysis, defined as presence of elevated methylcitric acid and no evidence of biotin related disorders in the organic acid analysis OR
  4. Diagnosed, or sibling diagnosed with MMA by semi-quantitative urine organic acid analysis, defined as elevation of methylmalonic acid and no evidence of vitamin B12 dependent disorder on plasma amino acid analysis
* Able to receive medications orally, by nasogastric (NG)-tube or by gastric (G)-tube
* No concomitant illness which would preclude safe participation as judged by the investigator
* Signed informed consent by the subject's legally acceptable representative
* After initial enrollment, criteria 3 or 4 (definitive diagnosis of the patient) must be fulfilled prior to discharge from initial admission in order to remain in the study.

Exclusion Criteria

* Had any prior hyperammonemic episode
* Administration of NCG within 7 days of participation in the study
* Use of any other investigational drug, biologic, or therapy, with the exception of sodium benzoate or sodium phenylacetate if the latter were administered prior to diagnosis by acylcarnitine analysis (diagnostic inclusion criterion 2), or organic acid analysis (diagnostic inclusion criteria 3 & 4)
* Planned participation in any other clinical trial
* Diagnosis of any medical condition causing hyperammonemia which is not PA or MMA.
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the investigator, may put the subject at an additional risk by participating in this study
* Had a liver transplant or is scheduled for a liver transplant
* Is not expected to be compliant with this study in terms of returning to site for subsequent episodes of hyperammonemia crises or for long-term follow-up

Ages: 1 Hour to 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mendel Tuchman, MD, Principal Investigator — Children's National Research Institute
Locations (7):
- United States (7):
  - University of California Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - The Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital Boston, Boston, Massachusetts
  - University Hospitals of Cleveland/Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
A single participant was enrolled before the study closed. There are no analyses and if data are shared, this may compromise the confidentiality of this single participant from a very rare disease.

RESULTS

PARTICIPANT FLOW:
Groups:
- Carbaglu: Active NCG & Standard of Care
  N-carbamylglutamate: Active NCG & Standard of Care Chemical Composition: N-carbamyl-L-glutamic acid (NCG) The daily dose will be 100 mg/kg/ day. The doses are to be divided into 2 equal doses and administered orally or enterally by nasogastric or gastrostomy tube (standard of care will prevail when choosing the mode of drug administration).
  The tablets must be dispersed in a minimum of 2.5-10 ml of water and ingested immediately or administered by fast push through a syringe via a nasogastric or gastrostomy tube. The suspension has a slightly acidic taste.
  This drug will be administered for 7 days after admission or until discharge (whichever is sooner).
  Standard of Care: Standard of Care
Period: Overall Study
Arm/Group | Carbaglu | Placebo
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: One participant, infant under 1 month old, with organic acidemia.
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbaglu | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 |  | 1
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 4 (0) |  | 4 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
NH3 [Mean (Standard Deviation); unit: mcmol/L] | 223 (0) |  | 223 (0)

OUTCOME MEASURES:

1. Primary Outcome: Neurodevelopment
Description: Neurodevelopmental outcome as measured by Cognitive Composite (Bayley III), Motor Composite (Bayley III) and Functional Status Scale and safety of NCG treatment as measured by adverse events and laboratory blood tests
Time Frame: 30 months
Population: The study was closed prematurely. There is no analysis population.
Arm/Group | Carbaglu | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety is measured by tracking and detailing the number and type of adverse events and their severity based on the CTCAE.
Time Frame: Start of episode through 7 days or discharge (if earlier)
Measure: Number; unit: Participants
Arm/Group | Carbaglu | Placebo
Number analyzed (Participants) | 1 | 0
Participants | 1 |

ADVERSE EVENTS:
Arm/Group | Carbaglu | Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carbaglu (N=1) | Placebo (N=0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) — Mildly lethargic
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — tachypnea, hyperpnea
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — vomited early in the AM
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — large ketones in urine
Acidosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — serum bicarbonate abnormal
low white blood counts (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Low overall white blood counts and low absolute neutrophil count
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — low hemoglobin and hematocrit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No